CLINICAL TRIAL: NCT06747364
Title: Phosphatidylethanol and Other Ethanol Consumption Markers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Nathalie Hill-Kapturczak, Associate Professor, The University of Texas Health Science Center at San Antonio
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00000887; R01AA022361 (NIH)
Record Dates: First submitted 2024-12-18; First posted 2024-12-24 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Healthy Volunteer; Alcohol Consumption
Keywords: Healthy adult; Light, moderate and heavy drinkers
MeSH Terms: conditions — Alcohol Drinking; Lymphoma, Follicular | interventions — Ethanol

STUDY DESIGN:
Intervention Model Description: The alcohol administration study will occur at the Applied Physiology Laboratory (APL) at UNT. The naturalistic drinking study will occur at UNT and a 2nd cohort will undergo a naturalistic drinking study at UTHSCSA Behavioral Research Lab (BRL).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- In Lab alcohol consumption followed by 10 days of abstinence and then 28-days naturalistic drinking (Experimental): Up to 40 Healthy volunteers will consume alcohol in the lab designed to produce a peak blood alcohol concentration of 0.06% and have blood collected over 6 hours. Followed by 10 days of abstinence and 4 visits to provide 1 blood sample each time. These 40 participants will then consume alcohol as usual outside the laboratory for 28 days and blood will be collected weekly (Day 0, Day 7, Day 14, 21 and 28). A second cohort of 40 participants will then undergo the naturalistic portion with blood collected on Days 0, Day 7, Day 14, 21 and 28.
  Interventions: Other: Alcohol (Ethanol)

INTERVENTIONS:
Other: Alcohol (Ethanol) — Alcohol will be administered to participants by research staff. In Phase 1, participants will consume alcohol designed to produce a targeted blood alcohol concentration (BAC) of 0.06% using the modified Widmark equation.

SUMMARY:
This study is intended to help the investigators understand how a biomarker found in the blood may be used to better identify the quantity and different patterns of alcohol use.

The investigators hope that the results of this study will help identify the uses of alcohol-use markers in the blood in future alcohol prevention and treatment programs. It is hoped that the information learned from this study will benefit other people in the future.

The study participants will come into the lab and will (1) consume alcohol in the lab designed to produce a peak blood alcohol concentration of 0.06% and have blood collected over 6 hours followed by abstinence for 10 days to give a small blood sample 4 times and (2) to give a small amount of blood 5 times within 28 days (naturalistic drinking) and provide answers about alcohol use.

DETAILED DESCRIPTION:
The study goal is to account for individual differences in biological variables likely influencing Phosphatidylethanol (PEth) formation to determine the extent to which the investigators can improve their ability to characterize alcohol consumed previously. Investigators propose three experiments that combine: (a) controlled human laboratory studies in vivo, (b) clinical laboratory studies of important enzymatic and biological variables measured ex vivo, and (c) the creation and testing of regression models to predict drinking during a naturalistic observational study using PEth levels and key biological variables identified in the lab.

Aim 1 is an in vivo pharmacokinetic study that whereby participants will consume a dose of alcohol to achieve a target blood alcohol concentration of 0.06%. Blood samples will be collected repeatedly during a 6-hour period to characterize blood/breath alcohol concentrations and PEth syntheses. Then PEth elimination half-life will be characterized across a 10-day period while remaining alcohol abstinent outside the lab.

In Aim 2, alcohol-free blood collected from Aim 1 will be examined ex vivo to characterize key biological variables (e.g., enzyme activity, red blood cell count, precursor levels) involved in PEth synthesis and elimination. Regression formulas will evaluate these variables for their ability to explain the previously unexplained between-subject differences in the PEth levels formed after the same amount of alcohol is consumed.

Finally, in Aim 3, regression equations will be used to evaluate the value of using these biological/enzyme variables to improve (above and beyond that of PEth alone) the prediction of naturalistic drinking self-reported by participants over a 28-day period.

ELIGIBILITY:
Inclusion Criteria:

1. are ≥ 21 years old;
2. are height and weight proportionate (body mass index 18-30); and
3. report drinking on > 1 days in the last month, with at least one day equal to at least achieving ~0.06% BAC.

Exclusion Criteria:

1. have significant current or predicted alcohol withdrawal symptoms (CIWA-AR scores ≥ 10);
2. are currently in alcohol treatment;
3. have substance use disorder (except nicotine, and/or caffeine);
4. have a medical condition that would contraindicate participation (a positive urine pregnancy test, self-reported scheduled surgery or liver disease);
5. are currently breast feeding;
6. have a presence of a DSM-5 psychiatric disorder with symptoms of psychosis and/or delirium; or
7. are unable to comprehend the informed consent process or study instructions.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-01-07 (Actual); Primary Completion 2029-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Phosphatidylethanol (PEth) concentrations on alcohol administration day in Males/Females | Baseline to 360 minutes
  Measure of PEth level in ng/ml over 360 minutes
Breath alcohol concentrations on alcohol administration day in Males/Females | Baseline to 360 minutes
  Measure of breath alcohol concentrations in g/dL over 360 minutes
PEth Concentrations for half-life in Males/Females | End of Day 0 to 10 days
  Measure of PEth concentrations in ng/ml on days 0 (end of day), 3, 5, 7 and 10
PEth concentrations once weekly during 28 days naturalistic drinking in Males/Females | Baseline to 28 days
  Measure of PEth level in ng/ml on days 0, 7, 14, 21 and 28
Self-reported drinking during the 28 days naturalistic drinking in Males/Females | Baseline to 28 days
  TLFB on days 0, 7, 14, 21 and 28
PEth Concentrations during the 28 days naturalistic drinking in Males/Females | Baseline to 28 days
  Measure of PEth concentrations in ng/ml on days 0, 7, 14, 21 and 28
Red blood cell count (RBC) in Males/Females | One time (baseline)]
  Measurement of RBCs in cells/mm^3
Phosphatidylcholine (PC) content in Males/Females | One time (baseline)
  Measurement of PC content in ng/ml at baseline
Ex vivo PEth formation for PLD activity in blood from Males/Females | Baseline to 90 minutes
  PEth concentrations in ng/mL at 0, 15, 30, 45, 60, and 90 min after alcohol exposure

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Hill-Kapturczak, PhD, Principal Investigator — The University of Texas Health Science Center at San Antonio; Donald Dougherty, PhD, Principal Investigator — University of North Texas Health Science Center
Locations (2):
- United States (2):
  - University of North Texas, Denton, Texas
  - University of Texas Health Science Center San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Public policy will focus on ensuring that all dissemination of deidentified individual participant research findings from this study is conducted in an accurate, transparent and ethical manner. Authorship will be determined based on significant contributions to the study's conception, design, data acquisition, analysis or interpretation as well as in drafting and critically revising the manuscript. All authors must approve the final version of the manuscript. The primary author will be the individual who has made the most significant contribution to the study, while co-authors will include those who have made substantial contributions.
  Final copies of all publications, abstracts, and presentations will be archived in the study's repository and made accessible to all study personnel, including the submitted version and any subsequent revisions.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: At the time of summary result reporting in ClinicalTrials.gov and when published in a peer review journal.